CLINICAL TRIAL: NCT04607304
Title: ABCA2 GIRMS Analytical Validation Clinical Performance Study - Patient Sample Collection
Brief Title: ABCA2 GIRMS Analytical Validation Clinical Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairn Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO-CD-044
Record Dates: First submitted 2020-10-18; First posted 2020-10-29 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Gastroparesis
Keywords: Gastroenterology; Gastric Emptying Breath Test
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ABCA2 GIRMS (Experimental): Leftover breath samples analyzed on ABCA2 GIRMS systems, order of analysis randomized
  Interventions: Device: ABCA2 GIRMS

INTERVENTIONS:
Device: ABCA2 GIRMS — Two systems (ABCA-C and ABCA-D) with run order randomized

SUMMARY:
The purpose of this study is to collect human breath samples for use in a validation study intended to demonstrate equivalent clinical performance measures of new ABCA2 GIRMS (Automated Breath Carbon Analyzer-2 Gas Isotope Ratio Mass Spectrometer) instruments to the currently FDA-approved ABCA GIRMS (Automated Breath Carbon Analyzer Gas Isotope Ratio Mass Spectrometer) system. ABCA GIRMS systems are used to analyze the ratio of 13CO2 to 12CO2 in patient breath samples during the GEBT (Gastric Emptying Breath Test) procedure.

DETAILED DESCRIPTION:
In this study the participants will be administered the FDA-approved GEBT test, which involves collecting breath samples prior to and after consumption of a non-radioactive carbon stable isotope (13C) labeled test meal. Breath samples will be collected at times consistent with FDA approved labeling. Participant's breath samples will be analyzed on the currently approved ABCA GIRMS and on the new ABCA2 GIRMS instruments. The values collected from both systems will be used to determine the clinical diagnostic agreement at each individual time points and percent agreement in diagnosis between the approved ABCA GIRMS and the new ABCA2 GIRMS.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-85 old at time of signing the informed consent form fro healthy and intended use population participants (i.e. symptomology of gastroparesis). Women of childbearing potential must not be pregnant at the time of GEBT administration.
* Ability to eat test meal and provide breath samples

Exclusion Criteria:

* History or physical exam suggestive of pathophysiologic disorders such as renal failure, chronic heart disease, chronic respiratory disease, liver disease or malabsorption syndrome
* History of abdominal surgery except appendectomy
* Use of any medications that may alter gastric motility within two days of the study
* Use of narcotics or anticholinergics within two days of the study
* Females on hormone replacement therapy other than birth control medications
* Receipt of an investigational drug within 4 weeks of the study
* Pregnancy
* Intolerance or allergy to any component of Gastric Emptying Breath Test meal
* History of neurologic or psychiatric disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Diagnostic agreement at each individual timepoints | Up to 7 days per participant
  Gastric emptying rates (kPCD) values compared between the validated ABCA GIRMS system and the new ABCA2 GIRMS systems for each GEBT post meal collection timepoint (45, 90, 120, 150, 180 and 240-minute timepoints) and the overall diagnosis
Percent agreement in diagnosis | Up to 7 days per participant
  Diagnosis compared between the comparative method (ABCA GIRMS) and the candidate method (ABCA2 GIRMS) at each post meal timepoint and the overall diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Alex Ryder, MD, Principal Investigator — Cairn Diagnostics
Locations (1):
- Cairn Diagnostics, Brentwood, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT04607304/Prot_SAP_000.pdf